CLINICAL TRIAL: NCT02826655
Title: Adaptive Optics for Ophthalmic Technologies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00071278
Record Dates: First submitted 2016-07-01; First posted 2016-07-11 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: WF-OCT; OCT; diabetic retinopathy; diabetic macular edema
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Controls (Active Comparator): Study participants will undergo imaging of both eyes with the WF-AO-OCT unit, per standard operating protocol. Imaging is noncontact. Study participants will undergo only a single imaging session on a single day.
  Interventions: Device: WF-AO-OCT
- Subjects with diabetic retinopathy (Experimental): Study participants will undergo imaging of both eyes with the WF-AO-OCT unit, per standard operating protocol. Imaging is noncontact. Study participants will undergo only a single imaging session on a single day.
  Interventions: Device: WF-AO-OCT

INTERVENTIONS:
Device: WF-AO-OCT — WF-AO-OCT allows noninvasive, high-resolution imaging of the microvasculature of the retina and choroid, without intravenous dye administration. This unit is being conducted under an abbreviated IDE.

SUMMARY:
This is a feasibility study to assess the use of wide field adaptive optics optical coherence tomography (WF-AO-OCT) to determine whether there are structural differences in the peripheral retina in participants diagnosed with diabetic retinopathy compared to a healthy control group. This study being conducted under an abbreviated IDE. The investigators will analyze data using descriptive statistics. Risks related to light exposure will be managed by ensuring that the exposure to the WF-AO-OCT light source is well below maximum permissible limits for safe exposure.

DETAILED DESCRIPTION:
Adaptive optics (AO) is an optical technique that corrects the natural aberrations (optical imperfections) of the eye. Since it was first described in 1997, it has been used successfully to enhance the visualization of retinal tissue, in particular, the human photoreceptor mosaic. Previous studies using AO in the human eye have contributed to considerable advancements in our understanding of vision and ocular pathologies.

An AO system sends a pattern of light into the eye that balances the eye's inherent imperfections. This leads to better imaging by providing better light focusing by the natural lens of the eye. The AO system measures the light returning from the eye as is typical in clinically accepted optical coherence tomography and scanning laser ophthalmoscope systems.

A schematic AO system consists of a light input, a deformable/adaptive mirror that modifies the shape of the light entering and exiting the eye, and a detector system that captures and analyzes the returning light from the eye.

The device used in this feasibility study has been tested to ensure that its light output is within ANSI limits for safe ocular exposure and is capable of obtaining useful images of the peripheral retina in normal subjects.

Diabetic retinopathy represents the most common cause of vision loss in working aged adults. Vision loss is related to two manifestations of advanced diabetic retinopathy: proliferative diabetic retinopathy (PDR) and diabetic macular edema (DME). PDR occurs when the vascular perfusion of the retina is compromised and compensatory signals including expression of vascular endothelial growth factor causes neovascularization on the surface of the retina. These abnormal vessels cause vision loss by either bleeding into the vitreous or by contracting leading to retinal detachment. DME occurs when vascular leakage results in swelling of the macular tissue causing central vision loss. While DME affects the macula (the area typically imaged using OCT), PDR is much more frequently found in the peripheral retina which is not typically imaged by traditional OCT devices. In recently years, wide field fluorescein angiography has allowed insights into the relationship between DME, PDR and the status of retinal blood vessels within the macula and the retinal periphery. WF-AO-OCT has the potential to provide similar or complementary structural detail of the retinal tissue and vasculature within the macula and retinal periphery. The advantage of WF-AO-OCT is that it is a non-contact, non-invasive imaging technology which is easier to use, faster and less invasive compared to fluorescein angiography which entails intravenous injection of fluorescein, requires a skilled ophthalmic photographer and takes 10-20 minutes to perform. By imaging participants who have previously undergone wide field fluorescein angiography as standard of care, the investigators will be able to compare the information obtained using WF-AO-OCT and to determine its sensitivity in identifying specific vascular and morphological findings associated with PDR and DME.

ELIGIBILITY:
Inclusion Criteria for diabetic retinopathy participants:

* Diagnosis of diabetic retinopathy in one or both eyes
* Men and Women, aged 18 years or older
* Able to provide written informed consent

Inclusion Criteria for healthy control participants:

* No history of retinal disease in one or both eyes
* Men and Women, aged 18 years or older
* Able to provide written informed consent

Exclusion Criteria for both diabetic retinopathy and healthy control participants:

* Significant media opacity (e.g. cataract or vitreous hemorrhage) precluding clinical imaging adequate for interpretation
* Unwilling or unable to provide legally effective written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Image Quality | 30 minutes
  Assessment of quality of images obtained by WF-AO-OCT unit.
Peripheral Retina Structure Differences between Healthy Controls and participants with diabetic retinopathy. | 30 minutes
  Differences between the control and case populations will be described using descriptive statistics. This data can then be used to power future, more dedicated studies.

CONTACTS AND LOCATIONS:
Overall Officials: Sina Farsiu, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States